CLINICAL TRIAL: NCT01949857
Title: Phase 4 Clinical Trial to Assess the Safety, Immunogenicity,Three-year Immune Persistence of Inactivated Hepatitis A Vaccine (HAV) and Live Attenuated HAV Vaccine
Brief Title: The Immunogenicity and Safety of Inactivated and Live Attenuated Hepatitis A Vaccines
Acronym: HAV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: qiangmingsun123456!
Record Dates: First submitted 2013-08-28; First posted 2013-09-25 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Hepatitis A
Keywords: Hepatitis A; Vaccine; Safety; efficacy
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines; Vaccines; Freeze Drying

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Attenuated HAV Vaccine, H2 Strain (Experimental): 6.50 lgCCID50/ml in babies aged 18-35 months\6.50 lgCCID50/ml in children aged 3-15 years \6.50 lgCCID50/ml in adults aged 16 up to 65 years old
  Interventions: Biological: Attenuated HAV Vaccine, H2 Strain
- Attenuated HAV Vaccine, L-A-1 Strain (Experimental): 6.50 lgCCID50/Vial in babies aged 18-35 months\6.50 lgCCID50/Vial in children aged 3-15 years \6.50 lgCCID50/Vial in adults aged 16 up to 65 years old, only one dose (1Vial/dose).
  Interventions: Biological: Attenuated HAV Vaccine, L-A-1 Strain
- Inactivated HAV Vaccine, Lu8 Strain (Experimental): 320EU/Vial in babies aged 18-35 months\320EU/Vial in children aged 3-15 years \640EU/Vial in adults aged 16 up to 65 years old\boost at month 6\two-dose
  Interventions: Biological: Inactivated HAV Vaccine, Lu8 Strain
- Inactivated HAV Vaccine, TZ84 Strain (Experimental): 250U/Vial in babies aged 18-35 months\250U/Vial in children aged 3-15 years \500U/Vial in adults aged 16 up to 65 years old\boost at month 6\two-dose
  Interventions: Biological: Inactivated HAV Vaccine, TZ84 Strain

INTERVENTIONS:
Biological: Attenuated HAV Vaccine, H2 Strain — 6.50 lgCCID50/Vial in babies aged 18-35 months\6.50 lgCCID50/Vial in children aged 3-15 years \6.50 lgCCID50/Vial in adults aged 16 up to 65 years old, only one dose (1Vial/dose).
  Other Names: Hepatitis A (Live) Vaccine, Freeze-dried
  Arms: Attenuated HAV Vaccine, H2 Strain
Biological: Attenuated HAV Vaccine, L-A-1 Strain — 6.50 lgCCID50/Vial in babies aged 18-35 months\6.50 lgCCID50/Vial in children aged 3-15 years \6.50 lgCCID50/Vial in adults aged 16 up to 65 years old, only one dose (1Vial/dose).
  Other Names: Hepatitis A Vaccine
  Arms: Attenuated HAV Vaccine, L-A-1 Strain
Biological: Inactivated HAV Vaccine, Lu8 Strain — 320EU/Vial in babies aged 18-35 months\320EU/Vial in children aged 3-15 years \640EU/Vial in adults aged 16 up to 65 years old\boost at month 6\two-dose
  Other Names: Hepatitis A Vaccine, Inactivated
  Arms: Inactivated HAV Vaccine, Lu8 Strain
Biological: Inactivated HAV Vaccine, TZ84 Strain — 250U/Vial in babies aged 18-35 months\250U/Vial in children aged 3-15 years \500U/Vial in adults aged 16 up to 65 years old\boost at month 6\two-dose.
  Other Names: Hepatitis A Vaccine, Inactivated
  Arms: Inactivated HAV Vaccine, TZ84 Strain

SUMMARY:
The purpose of this Phase 4 trial is to assess the safety, immunogenicity, three-year immune persistence of inactivated hepatitis A vaccine (HAV) and live attenuated HAV vaccine.

DETAILED DESCRIPTION:
Hepatitis A refers to liver inflammation caused by infection with the hepatitis A virus. HAV is is one of the most common hepatitis viruses that can cause hepatitis in China. The data from the phase 1, 2 and 3 trials suggested that both inactivated hepatitis A vaccine and live attenuated hepatitis A vaccine had a clinically acceptable safety and good immunogenicity for healthy Chinese people.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects fulfilling all of the following criteria will be eligible for the study:

  * People aged from 18 months to 65 years old.
  * The subjects or subjects' guardians are able to understand and sign the informed consent
  * The subjects or subjects' guardians allow to comply with the requirements of the protocol
  * Subjects with temperature <=37.0°C on axillary setting
  * The subjects have signed informed consent already

Exclusion Criteria:

* Subjects will not be eligible for the study if any of the following criteria is met:

  * Subject who has a medical history of serious disease including Tumor, autoimmune disease, progressive atherosclerosis diseases or complications of diabetes, chronic obstructive pulmonary disease (copd), kidney disease, congestive heart failure etc.
  * Have a history of neurological symptoms or signs
  * Have medical history or family history relating to allergies, seizures, epilepsy, brain and spirit etc.
  * Suffering from serious chronic diseases
  * Suffering from known or suspected of diseases including respiratory diseases, acute infection , mothers have HIV infection, cardiovascular disease, severe hypertension, skin diseases, malignant tumor
  * Allergic to any ingredient in research, history of allergies to any vaccination (always), especially for people allergic to high protein food like eggs and milk
  * Any prior known or suspected damage or abnormal immune function. As for patients who are treated with immune inhibitors or immune enhancer medicine, accept with immunoglobin, blood products and plasma extraction within 3 months
  * Any prior diseases including human immunodeficiency virus infection or related
  * Bleeding constitution or prolong bleeding time situation
  * Accept hepatitis A vaccination within a month
  * Received vaccines, other immune globulin, any research drug injections in the past 4 weeks
  * People who had any acute illness, needed systemic antibiotics or antiviral treatment in the past 7 days
  * Caught a fever with axillary temperature 38°C or higher in past 3 days
  * Take part in another clinical researchers
  * Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
  * Pregnancy test result is positive

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35000 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
changes of hepatitis A antibody concentration | up to 43 months
  1. Changes of anti-HAV antibody geometric mean concentrations at pre-vaccination, month 1,12, 24, 36, and 1 months after the booster vaccination.

SECONDARY OUTCOMES:
The frequency of all the adverse events in vaccine group and placebo group | up to 43 months
  compare frequency of all the solicited events, unsolicited adverse events and serious adverse events between vaccine group and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Qihan Li, Ph.D., Study Chair — Institude of Medical Biology, Chinese Academy of Medical Sciences; Jingsi Yang, Study Chair — Institude of Medical Biology, Chinese Academy of Medical Sciences; Qiangming Sun, Ph.D., Principal Investigator — Institude of Medical Biology, Chinese Academy of Medical Sciences; Fubao Ma, Study Director — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Institute of Medical Biology -Chinese Academy of Medical Sciences, Kunming, Yunnan, China